CLINICAL TRIAL: NCT05366595
Title: Zinc Supplementation in Pediatric Sepsis; a Randomized Controlled Trial
Brief Title: Zinc Supplementation in Pediatric Sepsis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amal Osman, Assistant professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.19.05.614
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2022-05

CONDITIONS: Zinc in Pediatric Sepsis
MeSH Terms: interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): who received oral zinc sulfate supplementation on dose doses ranging from 10 mg (infants) to 20 mg (under-five children) of elemental zinc per day, a dosage that is safe in these children
  Interventions: Drug: oral zinc sulfate
- Control group (No Intervention): who didn't receive zinc sulfate supplementation.

INTERVENTIONS:
Drug: oral zinc sulfate — Oral zinc sulfate at dose 10 to 20 mg daily for 10 days
  Arms: Treatment group

SUMMARY:
a single blinded randomized controlled clinical trial that was conducted to evaluate the role of zinc supplementation in improving the outcome of infants and children with sepsis in pediatric intensive care unit.

DETAILED DESCRIPTION:
a single blinded randomized controlled clinical trial that was conducted to evaluate the role of zinc supplementation in improving the outcome of infants and children with sepsis in pediatric intensive care unit.

The study included 72 cases that were randomly divided into 2 groups

A- Group A (Zinc treated group):

Included 36 cases who received oral zinc sulfate supplementation at doses ranging from 10 mg (infants) to 20 mg (under-five children) of elemental zinc per day, a dosage that is safe in these children.

B- Group B:

Included 36 cases who didn't receive zinc sulfate supplementation.

Method of randomization:

The cases were randomly divided into two groups using the closed envelope technique. The numbers from 1 to 72 were written in flat pieces of papers and put in closed envelopes that were randomly distributed to the participants.

The cases with the odds number were allocated to the zinc treated group while the cases with the even numbers were allocated to the other group.

ELIGIBILITY:
Inclusion Criteria:

* 2- Pediatric patients who fulfill Pediatric Consensus criteria for definition of severe sepsis as 1) greater than or equal to 2 age-based systemic inflammatory response syndrome criteria, 2) confirmed or suspected invasive infection, and 3) cardiovascular dysfunction, acute respiratory distress syndrome, or greater than or equal to 2 organ system dysfunctions

Exclusion Criteria:

* Infants and children with history of prematurity (< 37 weeks), chronic cardiopulmonary disease, immunodeficiency, neuromuscular disease, surgical conditions and any other chronic medical condition.
* Those who are regularly taking vitamin or mineral supplementations

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Mortality rate | through study completion an average of one year
  Frequency of occurrence of death

SECONDARY OUTCOMES:
Zinc level | after 10 days of treatment
  serum zinc level

CONTACTS AND LOCATIONS:
Overall Officials: Angi A Al Wakil, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University Children's Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Results will be published by the investigators in academic journals. Sharing of generated study data will be carried out in several different ways. We plan to make our results available to researchers and potential interested collaborators